CLINICAL TRIAL: NCT06960915
Title: Efficacy of Virtual Reality Reminiscence Therapy in Nursing Home Residents With Alzheimer's Disease or Related Diseases
Acronym: ReminiSOMME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PI2025_843_0068
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Virtual Reality; Reminiscence Therapy; Nursing Home; Alzheimer's Disease or Related Diseases; Crossover Study
Keywords: Virtual reality; Reminiscence therapy; Nursing home; Alzheimer's disease or related diseases; crossover study

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immersive virtual reality (Experimental): The residents will be equipped with a virtual reality headset where they will enjoy 360° panoramas that will immerse them in the heart of villages in the Amiens basin and in particular their village based on 3 to 5 images per village: church square, village square, town hall, emblematic places, etc
  Interventions: Device: immersive virtual reality
- classic reminiscence workshops (Active Comparator): classic reminiscence workshops in which the organizer will propose to discuss memories and past experiences using photographs, objects or music in the control arm
  Interventions: Device: classic reminiscence workshops

INTERVENTIONS:
Device: immersive virtual reality — The research procedure will be the realization of reminiscence workshops in immersive virtual reality. The residents will be equipped with a virtual reality headset where they will enjoy 360° panoramas that will immerse them in the heart of villages in the Amiens basin and in particular their village based on 3 to 5 images per village: church square, village square, town hall, emblematic places, etc.
  Arms: immersive virtual reality
Device: classic reminiscence workshops — It will be compared to classic reminiscence workshops in which the organizer will propose to discuss memories and past experiences using photographs, objects or music in the control arm.
  Arms: classic reminiscence workshops

SUMMARY:
This project provides the easiest possible access to heritage elements that older persons with Alzheimer's disease or related diseases knew well but to which they no longer have access due to the motor and functional dependencies they present. It will strengthen the possibilities of reminiscence by using, rather than the usual supports, virtual reality technology to reinforce the immersion effect. It will involve carrying out virtual reality reminiscence workshops intended for residents in nursing home with Alzheimer's disease or related diseases and allowing them to explore the heritage of towns and villages in the Somme region thanks to these innovative solutions. The aim of this project is to reduce behavioral disorders and improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Residents of the long-term care facilities of the Amiens-Picardie University Hospital,
* Residents with mild to moderate Alzheimer's disease or related diseases, i.e. with an MMSE ≥ 10,
* Residents or their legal representative agreeing to participate in the study.

Exclusion Criteria:

* Non-residents of the long-term care facilities of the Amiens-Picardie University Hospital,
* Residents with an MMS < 10,
* Residents or their legal representative refusing to participate in the study,
* Residents in terminal palliative care,
* Residents with disruptive behavioral disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Reduced behavioral problem frequency in immersive virtual reality group | 1 year
  Efficacy in reducing behavioral problems will be assessed using the sum of scores on the NPI-ES anxiety, depression, and apathy subscales.

SECONDARY OUTCOMES:
Improved quality of life in the immersive virtual reality group | 1 year
  improving the quality of life will be assessed using a quality of life scale developed for patients with Alzheimer's disease or related diseases, the QOL-AD scale validated in French.
  The QOL-AD is administered in interview format to individuals with dementia, following the instructions below.
  Scoring instructions for QOL-AD:
  Points are assigned to each item as follows: poor = 1, fair = 2, good = 3, excellent = 4.
  The total score is the sum of all 13 items.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No